CLINICAL TRIAL: NCT00959439
Title: A Comparative Bioavailability Study of Naproxen Delayed-Release Tablets, 375mg.
Brief Title: Relative Bioavailability Study of Naproxen Delayed-Release Tablets (375 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11704
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis | interventions — Naproxen

ARMS (2):
- 1 (Experimental): Naproxen Delayed Release Tables, 375 (Gevena Pharmaceuticals, Inc.)
  Interventions: Drug: Naproxen Delayed Release Tables, 375 (Gevena Pharmaceuticals, Inc.)
- 2 (Active Comparator): Naproxen (EC-Narosyn) Delayed Release Tables, 375 (Syntex (USA), Inc.)
  Interventions: Drug: Naproxen (EC-Narosyn) Delayed Release Tables, 375 (Syntex (USA), Inc.)

INTERVENTIONS:
Drug: Naproxen Delayed Release Tables, 375 (Gevena Pharmaceuticals, Inc.)
  Arms: 1
Drug: Naproxen (EC-Narosyn) Delayed Release Tables, 375 (Syntex (USA), Inc.)
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioavailability of Naproxen delayed-release tablets (375 mg).

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2002-03; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 55 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.